CLINICAL TRIAL: NCT02955979
Title: Incidence of Acute Renal Failure Associated With Iodinated Contrast Agents in Pediatrics. Study CANOPY. Prospective Multicenter Study
Brief Title: Incidence of Acute Renal Failure Associated With Iodinated Contrast Agents in Pediatrics
Acronym: CANOPY
Status: Terminated | Type: Observational
Why Stopped: Due to lack of funding
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1608041; Y6D1846194a (Registry Identifier: CNIL); 16-532bis (Other: CCTIRS)
Record Dates: First submitted 2016-10-26; First posted 2016-11-04 (Estimated); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Acute Renal Insufficiency
Keywords: acute renal insufficiency; Iodinated Contrast Agents; pediatric
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CT scan with iodinated contrast agents: Patients under 16 years old and must pass a CT scan with iodinated contrast agents. The following data will be collected in the medical record (creatinine prior to injection, comorbidities and child characteristics, associated treatments and risk factors of acute renal failure, as well as the injection pattern).
  Interventions: Other: CT scan with iodinated contrast agents

INTERVENTIONS:
Other: CT scan with iodinated contrast agents — Before the CT scan, the investigators with iodinated contrast agents, the following data will be collected in the medical record: creatinine prior to injection, comorbidities and child characteristics, associated treatments and risk factors of acute renal failure, as well as the injection pattern.
  After the CT scan the investigators will collect the characteristics of the injection type, osmolarity and volume of contrast used and the appearance of a possible allergic reaction.
  Then 24 and 48 hours and day 7 will collect serum creatinine, urine output and vital replacement therapies may be necessary.

SUMMARY:
Iodinated contrast media are now frequently used in diagnostic imaging exams, including pediatrics.

In adults, the acute renal failure (ARF) associated with contrast agents (CA-AKI) occur in 3-33% of exposed patients, especially as the patient is fragile, has comorbidities or pre-existing renal aggression .

In children, the prevalence of this little known disease is probably underestimated.

The investigators intend to conduct a prospective epidemiological study, to estimate the impact of the acute renale failure to iodinated contrast agents in pediatrics.

DETAILED DESCRIPTION:
Patients will be included those of pediatric emergencies, Hospitalization Unit of Short Duration pediatric, pediatric intensive care and pediatric resuscitation. The acute renale failure will be estimated on the basis of criteria KDIGO (score of kidney disease) group in 2012 to 48 hours a computed tomography (CT) scan with injection of contrast media, based on a change in creatinine clearance of the estimated according to the formula Schwartz revised in 2009 and / or diuresis.

Patient characteristics will be identified in order to establish risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients under 16 years admitted to a participating service
* Patient receiving an injected CT scan

Exclusion Criteria:

* Prior Inclusion in the study during an earlier review.
* Opposition of parents.
* Chronic renal failure or end-stage requiring renal replacement in the long term.

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: patients less than 16 years and who enjoys receiving an injected CT.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Creatinine | change from baseline creatinine at 7 days
  data gathered in the medical file
Diuresis | change from baseline diuresis at 7 days
  data gathered in the medical file

SECONDARY OUTCOMES:
Readmission | at 7 days
  Number of patients with no or having an adverse event during the readmission.
Hospitalization in intensive care | at 7 days
  Number of patients with no or having an adverse event during the hospitalization in intensive care.
Renal replacement | at 7 days
  Number of patients with no or having an adverse event during the renal replacement.
Death | at 7 days
  Number of dead

CONTACTS AND LOCATIONS:
Overall Officials: Olivier MORY, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (2):
- France (2):
  - CHU de Lyon, Lyon
  - Chu Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No